CLINICAL TRIAL: NCT01841047
Title: Assessment of Helical Tomotherapy Radiotherapy (54 Gy) Followed by Surgery in Retro-peritoneal Liposarcoma
Acronym: TOMOREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2008-42
Record Dates: First submitted 2012-11-05; First posted 2013-04-26 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2021-02

CONDITIONS: Liposarcoma
Keywords: Retroperitoneal liposarcoma operable
MeSH Terms: conditions — Liposarcoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Other): Evaluation of the combination of radiotherapy with helical tomotherapy (54 Gy) followed by surgery in retro-peritoneal liposarcomas.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Evaluation of the efficacy of the combination with radio-surgery helical tomotherapy irradiation to a dose of radiation of 54 Gy in patients with retroperitoneal liposarcoma of operable

SUMMARY:
Retro peritoneal liposarcomas are rare (less than 15% of sarcomas) whose prognosis is locoregional.

In the treatment of retroperitoneal liposarcomas main prognostic factor is the quality of the surgical resection. The effect of radiotherapy combined with surgery is uncertain and until now limited perhaps because of limited prescribed doses (of the order of 45Gy to 50Gy) due to high risk of organ toxicity nearby.

The helical tomotherapy is an innovative equipment radiotherapy to make conformational radiotherapy modulation intensity and is particularly suitable for irradiations precision (imaging mode associated with daily scanner) in large complex volumes. Increasing doses (increase of the prescribed dose to 54 Gy, thus potentially curative), the helical tomotherapy should allow to improve the efficacy of radiotherapy.

DETAILED DESCRIPTION:
Retro peritoneal liposarcomas are rare (less than 15% of sarcomas) whose prognosis is locoregional. In the treatment of retroperitoneal liposarcomas main prognostic factor is the quality of the surgical resection. The effect of radiotherapy combined with surgery is uncertain and until now limited perhaps because of limited prescribed doses (of the order of 45Gy to 50Gy) due to high risk of organ toxicity nearby.

Two elements can overcome these difficulties:

* Preoperative radiotherapy made rather than Postoperatively, the tumor in place back the gastrointestinal tract and reducing toxicity,
* The contribution of conformal radiotherapy techniques with intensity modulation (IMRT). The helical tomotherapy is an innovative equipment radiotherapy to make conformational radiotherapy modulation intensity and is particularly suitable for irradiations precision (imaging mode associated with daily scanner) in large complex volumes. Increasing doses (increase of the prescribed dose to 54 Gy, thus potentially curative), the helical tomotherapy should allow to improve the efficacy of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Liposarcoma histologically proven, in case of non-contributive biopsy: diagnosis radiologically validated within a multidisciplinary meeting
2. Protocol TOMOREP technically feasible,
3. Patients over 18 years
4. Considered as resectable even if multi-visceral excision is needed
5. Absence of morbidity contra-indicating surgery. The evaluation will be performed by the surgeon or the radiotherapist according to the definitions by the ASA classification.
6. Original form (as well as tumors made after first incomplete excision) and form in first relapse.
7. Life expectancy greater than 6 months
8. Patient signed informed consent,
9. Patient affiliated to a social security.

Exclusion Criteria:

1. Metastasis associated
2. Extension intraperitoneal associated, mesenteric extension
3. bilaterally
4. Against disease-indicating the need for surgery (ASA 3 and 4).
5. Contra-indication to radiotherapy (such as prior radiotherapy into the volume to treat).
6. Patient included in another clinical trial
7. Patient unable to undergo medical monitoring test for any geographical, social or psychological reasons,
8. Private patient freedom and major subject of a measure of legal protection or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01-20 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KANTOR Guy, PU-PH, Study Chair — Institut Bergonié
Locations (5):
- France (5):
  - Centre Paul Strauss, Strasbourg, Alsace
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Claudius Regaud, Toulouse, Midi-Pyrénées
  - Centre René Gauducheau, Nantes, Pays de la Loire Region
  - Institut Curie, Paris, Île-de-France Region

REFERENCES:
- [Background] Sargos P, Stoeckle E, Ducassou A, Giraud A, Mervoyer A, Italiano A, Albert S, Ferron G, Bellera C, Kantor G. High dose (54 Gy) pre-operative helical tomotherapy for retroperitoneal liposarcoma: Results of a phase II multicenter study. Radiother Oncol. 2023 Sep;186:109791. doi: 10.1016/j.radonc.2023.109791. Epub 2023 Jul 10. PMID 37437608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 recruitment centers :
  * Institut Bergonié - Bordeaux
  * Claudius Régaud - Toulouse
  * René Gauducheau - Nantes
Groups:
- Radiotherapy: Evaluation of the combination of radiotherapy with helical tomotherapy (54 Gy) followed by surgery in retro-peritoneal liposarcomas.
  Helical tomotherapy (54 Gy) will take place over 6 consecutive weeks with 30 fractions of 1.8 Gy : 5 fractions per week followed by 2 days off. The surgery takes place between 2 and 8 weeks after the end of the tomotherapy.
Period: Overall Study
Arm/Group | Radiotherapy
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 63.1 [35.5 to 82.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26
Region of Enrollment [Number; unit: participants]
  France | 48
WHO status [Count of Participants; unit: Participants] — The WHO performance status classification categorises patients as:
  0: able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. symptomatic and in a chair or in bed for greater than 50% of the day but not bedridden
  4. completely disabled; cannot carry out any self-care; totally confined to bed or chair. Population: 1 patient with data not available
  Participants
    number analyzed (Participants) | 47
    0 | 31
    1 | 13
    2 | 2
    3 | 1
    4 | 0
Histotype [Count of Participants; unit: Participants] — Sub histological type of liposarcoma
  Participants
    Liposarcoma well differentiated | 20
    Liposarcoma dedifferentiated or pleomorphic | 28

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence Rate of Local Recurrence and Competing Risks (All Patients)
Description: Evaluation of the efficacy of the combination with radio-surgery helical tomotherapy irradiation to a dose of radiation of 54 Gy in patients with retroperitoneal liposarcoma of operable.
  The effectiveness will be evaluated in terms of local recurrence-free survival 3 years. Given the data and the lack of independence between local recurrence and metastasis events, the Kaplan Meier method cannot be applied. An estimation method adapted to the presence of competing risks is necessary. Including other events (metastasis, deaths...) consist in using a competing risk analysis methodology where the specific incidence of each type of event is estimated in the presence of the other types of events. The following results represent the cumulative incidence (as a percentage) of local recurrence on the one hand and the cumulative incidence of competing risks (distant metastasis or death) on the other hand.
Time Frame: 3 years from start of the tomotherapy treatment
Population: All patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 48
percentage of participants
  Cumulative incidence rate of local recurrence | 16.89 [7.90 to 28.75]
  Cumulative incidence rate of competing risks | 10.42 [3.82 to 20.86]

2. Primary Outcome: Cumulative Incidence Rate of Local Recurrence and Competing Risks (Liposarcoma Well Differentiated)
Description: Evaluation of the efficacy of the combination with radio-surgery helical tomotherapy irradiation to a dose of radiation of 54 Gy in patients with retroperitoneal liposarcoma of operable.
  The effectiveness will be evaluated in terms of local recurrence-free survival 3 years.Given the data and the lack of independence between local recurrence and metastasis events, the Kaplan Meier method cannot be applied. An estimation method adapted to the presence of competing risks is necessary. Including other events (metastasis, deaths...) consist in using a competing risk analysis methodology where the specific incidence of each type of event is estimated in the presence of the other types of events. The following results represent the cumulative incidence (as a percentage) of local recurrence on the one hand and the cumulative incidence of competing risks (distant metastasis or death) on the other hand.
Time Frame: 3 years from start of the tomotherapy treatment
Population: Analysis for the 20 patients with well-differentiated liposarcoma
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 20
percentage of participants
  Cumulative incidence rate of local recurrence | 5.00 [0.35 to 20.53]
  Cumulative incidence rate of competing risks | 5.00 [0.35 to 20.53]

3. Primary Outcome: Cumulative Incidence Rate of Local Recurrence and Competing Risks (Liposarcoma Dedifferentiated or Pleomorphic)
Description: as for outcome 2
Time Frame: 3 years from start of the tomotherapy treatment
Population: Analysis for the 28 patients with dedifferentiated or pleomorphic liposarcoma
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 28
percentage of participants
  Cumulative incidence rate of local recurrence | 25.71 [11.36 to 42.82]
  Cumulative incidence rate of competing risks | 14.29 [4.50 to 29.50]

4. Secondary Outcome: Percentage of Participants With Disease-Free Survival (All Patients)
Description: Evaluation of the efficacy of the combination with radio-surgery helical tomotherapy irradiation to a dose of radiation of 54 Gy in patients with retroperitoneal liposarcoma of operable.
  The effectiveness will be evaluated in terms of disease free survival rate at 3 years, with the kaplan-meier method.
  The disease-free survival time is calculated between the date of the start of the tomotherapy treatment and the date of death, distant metastasis or local recurrence (events), whichever occur first, or the date of last news (censorship).
Time Frame: 3 years from start of the tomotherapy treatment
Population: All patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 48
percentage of participants | 72.70 [57.65 to 83.14]

5. Secondary Outcome: Percentage of Participants With Disease-Free Survival (Liposarcoma Well Differentiated)
Description: as for outcome 4
Time Frame: 3 years from start of the tomotherapy treatment
Population: Analysis for the 20 patients with well-differentiated liposarcoma
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 20
percentage of participants | 90.00 [65.60 to 97.40]

6. Secondary Outcome: Percentage of Participants With Disease-Free Survival (Liposarcoma Dedifferentiated or Pleomorphic)
Description: as for outcome 4
Time Frame: 3 years from start of the tomotherapy treatment
Population: Analysis for the 28 patients with dedifferentiated or pleomorphic liposarcoma
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 28
percentage of participants | 60.00 [39.45 to 75.54]

7. Secondary Outcome: Percentage of Participants With Overall Survival (All Patients)
Description: Evaluation of the efficacy of the combination with radio-surgery helical tomotherapy irradiation to a dose of radiation of 54 Gy in patients with retroperitoneal liposarcoma of operable.
  The effectiveness will be evaluated in terms of overall survival rate at 1, 3 and 5 years, with the kaplan-meier method.
  The overall survival time is calculated between the date of the start of the tomotherapy treatment and the date of death (event), or the date of last news (censorship).
Time Frame: 1 year, 3 years and 5 years from start of the tomotherapy treatment
Population: All patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 48
percentage of participants
  1-year Overall survival rate | 93.62 [81.50 to 97.90]
  3-years Overall survival rate | 80.60 [66.02 to 89.40]
  5-years Overall survival rate | 73.94 [58.67 to 84.29]

ADVERSE EVENTS:
Time Frame: 5 years (all the study period for a patient, from date of inclusion to date of end of study)
Description: Only for SAEs were monitored/assessed. Other [Not Including Serious] Adverse Events were not monitored/assessed (so Total Number At Risk = 0).
Arm/Group | Radiotherapy
All-Cause Mortality (participants affected / at risk) | 13/48
Serious Adverse Events (participants affected / at risk) | 30/48
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy (N=48)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Disease progression (General disorders) | 8 (8)
Sudden death NOS (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Lymphocele (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes